CLINICAL TRIAL: NCT05288738
Title: Comparing Post-Operative Analgesic Effects of Patient-Controlled Analgesia Morphine (PCAM) in Combination With Dexmedetomidine 1 mcg/ml Versus PCAM With Dexmedetomidine 2 mcg/ml
Brief Title: Comparing Post-Operative Analgesic Effects of PCAM With Dexmedetomidine 1 mcg/ml vs PCAM With Dexmedetomidine 2 mcg/ml
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FF-2019-543
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2021-04

CONDITIONS: Post-Operative Analgesia; Opioid Use, Unspecified; Laparotomy Surgery
Keywords: PCA Morphine; Dexmedetomidine; Morphine-dexmedetomidine; PCA-adjunct
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D1 (Active Comparator): PCA morphine 1mg/ml
  Interventions: Drug: Dexmedetomidine 1 mcg/ml
- Group D2 (Active Comparator): PCA morphine 1mg/ml
  Interventions: Drug: Dexmedetomidine 2 mcg/ml

INTERVENTIONS:
Drug: Dexmedetomidine 1 mcg/ml — 34 patients received PCA morphine 1 mg/ml with combination of dexmedetomidine 1 mcg/ml
  Other Names: Precedex
  Arms: Group D1
Drug: Dexmedetomidine 2 mcg/ml — 34 patients received PCA morphine 1 mg/ml with combination of dexmedetomidine 2 mcg/ml
  Other Names: Precedex
  Arms: Group D2

SUMMARY:
PCA morphine have been a common method in providing excellent analgesia for post-operative period. However, the usage of morphine is not without any side effects such as nausea, vomiting, respiratory depression, and over sedation.

Many adjunct have been used in combination with morphine to observe the opioid sparing effects at the same time providing good analgesia.

Dexmedetomidine is a potent and selective alpha-2 receptor agonist with sedative, anxiolytic, sympatholytic, and analgesic effects. As dexmedetomidine and morphine act via different mechanism, this combination produces synergistic analgesic effects.

The objective of our study was to observe the effectiveness in pain relief between two low concentration of dexmedetomidine (2 mcg/ml versus 1 mcg/ml) as an adjunct to PCA morphine 1 mg/ml.

DETAILED DESCRIPTION:
This was a double-blinded prospective randomised study conducted in Universiti Kebangsaan Malaysia Medical Centre from January 2020 till November 2020. This study was approved by Dissertation Committee of the Department of Anaesthesiology and Intensive Care, Universiti Kebangsaan Malaysia Medical Centre (UKMMC) and Medical Research and Ethics Committee of UKMMC.

Consent was taken during preoperative visit whereby patients were counselled on the use of PCA machine and assessment of pain score using visual analogue scale (VAS). All patients were not given sedative premedication before surgery. Induction of general anaesthesia was with IV fentanyl 2 mcg/kg, IV propofol 2 mg/kg and paralysed with IV rocuronium 0.6 mg/kg. Patients were given IV dexamethasone 0.2 mg/kg for postoperative nausea and vomiting (PONV) prophylaxis. Anaesthesia was maintained with sevoflurane to achieve MAC of 1.0 with oxygen and air in 1:1 ratio. All patients received IV morphine 0.1mg/kg intraoperatively, and surgical site infiltrated with levobupivacaine 0.5% 2 mg/kg. IV granisetron 1 mg was given to all patients at the end of the surgery and reversal was with IV neostigmine 0.05 mg/kg and IV atropine 0.02 mg/kg.

All patients were connected to the PCA morphine with test drugs after arrival in the recovery area. Patients were encouraged to self-administer the PCA whenever required. In an event of uncontrolled pain, rescue analgesia was with IV fentanyl 20 mcg boluses. All patients upon discharged to ward from recovery bay must have pain score (VAS) of less than 4, respiratory rate more than 10, MAP > 65 mmHg and HR > 60 beats/minute.

Patients were followed up at 6, 12, and 24 hours after surgery to look at the cumulative PCA morphine usage, incidence of nausea and vomiting, sedation score, respiratory depression (respiratory rate < 10 breath/min/). Side effects from dexmedetomidine namely hypotension (MAP < 65) and bradycardia (HR < 60) were also documented. The severity of nausea and vomiting was defined as mild, moderate, or severe while sedation was assessed according to five levels: 0, 1, 2, 3 and 4.

The power calculation for this study was based on a pilot study observing PCA consumption in the first 24 hours after surgery, with a mean difference, 14.67 and pooled standard deviation 20.27 in regard to dosage delivered comparing PCA morphine with dexmedetomidine 1 mcg/ml to PCA morphine with dexmedetomidine 2 mcg/ml. A group of 34 subjects each would be needed for a study with an alpha level of 0.05 (two-tailed) and a beta level of 0.2 (80% power) including 10% dropout rate.

Data were analysed using IBMR SPSSRs Statistics MacOS version 26.0 (IBM Corporation, New York, United States of America). The results were presented as frequency (percentage) and standard deviation whenever appropriate. The cumulative PCA morphine and dexmedetomidine usage pain score was analysed using the Mann-Whitney U-test. The incidence of sedation and PONV was analysed using Chi-square. Heart rate and blood pressure were analysed using independent T-test. A probability level of < 0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 & 2 patient
* going for elective or emergency laparotomy surgery

Exclusion Criteria:

* patient with known allergy to morphine or dexmedetomidine
* Creatinine clearance less then 30ml/min
* Current alcohol dependency
* Psychiatric illness on regular sedative-hypnotic drugs
* significant obstructive sleep apnoea (OSA)
* Chronic pain patient who on regular opioids

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours
  Measure the total PCA morphine (mg) consumption post laparotomy

SECONDARY OUTCOMES:
Morphine side effects | at 6, 12, and 24 hours post laparotomy
  Assess the frequency and severity of morphine side effects with the use of PCA morphine post laparotomy (PONV, over sedation, respiratory depression)
Analgesic effects | at 6, 12, and 24 hours post laparotomy
  Assess patient's pain score post laparotomy
Dexmedetomidine side effects | at 6, 12, and 24 hours post laparotomy
  Assess frequency and severity of dexmedetomidine side effects (hypotension, bradycardia)

CONTACTS AND LOCATIONS:
Overall Officials: Yeoh Chih Nie, MMed, Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- Universiti Kebangsaan Malaysia Medical Center, Cheras, Kuala Lumpur, Malaysia